CLINICAL TRIAL: NCT05243303
Title: Augmenting Standard-of-care Treatment of Plaque Psoriasis by Neuromodulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burrell College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0090_2021
Record Dates: First submitted 2022-02-04; First posted 2022-02-17 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-04

CONDITIONS: Psoriasis Vulgaris
Keywords: transcutaneous auricular vagus nerve stimulation; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Patients with plaque psoriasis will be randomized in one of two groups: (1) Active treatment group. These patients will receive daily transcutaneous auricular vagus nerve stimulation for 3 months; (2) Control group. These patients will receive a sham procedure instead of the transcutaneous auricular vagus nerve stimulation.
Who Masked: Participant
Masking Description: Patients in both arms will not know in which of the two arms (active treatment or control group) they are randomized. The sham procedure is similar to the transcutaneous auricular vagus nerve stimulation (but does not involve the actual stimulation). Therefore, it is unlikely that patients are able to differentiate whether they are assigned to the control group or to the active treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active taVNS (Experimental): These patients will self-administer transcutaneous auricular vagus nerve stimulation (taVNS).
  Interventions: Device: Active taVNS
- Sham taVNS (Sham Comparator): These patients will self-administer a sham procedure mimicking the active taVNS procedure.
  Interventions: Device: Sham taVNS

INTERVENTIONS:
Device: Active taVNS — A bipolar clip electrode is placed at the cymba conchae of the ear. Through this bipolar clip electrode, afferent nerve fibers within the auricular branch of the vagus nerve will be stimulated. Subjects self-administer the stimulation on a daily basis for 3 months.
  Other Names: active transcutaneous auricular vagus nerve stimulation
  Arms: Active taVNS
Device: Sham taVNS — A bipolar clip electrode is placed at the cymba conchae of the ear. However, active stimulation of the afferent nerve fibers within the auricular branch of the vagus nerve will not occur, because the electrode wire is electrically interrupted. Subjects self-administer the sham taVNS on a daily basis for 3 months.
  Other Names: sham transcutaneous auricular vagus nerve stimulation
  Arms: Sham taVNS

SUMMARY:
The human body responds to inflammation, such as psoriatic skin lesions, by activating the cholinergic anti-inflammatory pathway. In patients with plaque psoriasis, this pathway is not sufficient to clear the skin lesions. Importantly, the vagus nerve, that is part of the anti-inflammatory pathway, also innervates the ear where it can be activated through non-invasive transcutaneous auricular vagus nerve stimulation (taVNS). This raises the research question if taVNS - added to standard of care - improves the symptoms of plaque psoriasis by augmenting the function of the cholinergic anti-inflammatory pathway. Thus, the aim of this project is to test the hypothesis that daily taVNS applied for 3 months results in anti-inflammatory actions and improvements in the Psoriasis Area and Severity Index (PASI). Potential anti-inflammatory actions of taVNS compared to a sham-taVNS control group will be assessed by plasma cytokine levels, flow cytometry, and cell culture experiments. This project is potentially significant, because it may demonstrate that taVNS lessens the symptoms of plaque psoriasis and, therefore, improves the quality of life of millions of patients.

DETAILED DESCRIPTION:
An estimated 20% of psoriasis patients experience treatment failure. Afferent vagal nerve fibers that are part of the anti-inflammatory reflex sense inflammation, such as psoriatic skin lesions. The investigators' pilot data show that transcutaneous auricular vagus nerve stimulation (taVNS) activates afferent nerve fibers within the auricular branch of the vagus nerve to trigger anti-inflammatory reflex responses in healthy individuals. However, it is unknown if taVNS improves plaque psoriasis through the anti-inflammatory reflex. The lack of studies on taVNS in plaque psoriasis constitutes a missed opportunity to reduce treatment failures.

The long-term goal of this research is to establish a neuromodulatory approach to activate the anti-inflammatory reflex in patients with plaque psoriasis to lessen treatment failures. The objective of this study is to test the hypothesis that taVNS elicits anti-inflammatory reflex responses and reduces the severity of plaque psoriasis.

In a single-blinded randomized controlled clinical trial, participants will self-administer taVNS or sham-taVNS (control) daily for a duration of 3 months, while continuing their standard-of-care treatment. At baseline, 7 days, and 1, 2, and 3 months, clinical , autonomic, and inflammatory responses will be assessed.

At the conclusion of this study, the investigators expect to demonstrate anti-inflammatory reflex responses to taVNS and reduced severity of plaque psoriasis. These outcomes are expected to have important positive impact, because they are anticipated to reduce treatment failures in patients with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Plaque psoriasis diagnosed by a dermatologist

Exclusion Criteria:

* pregnancy
* vestibulocochlear neuronitis or nerve damage
* cardiac arrhythmia
* epilepsy
* anticipated change in medication during the 3-month study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Psoriasis Area and Severity Index from Baseline at 1 Week | After 1 week of treatment.
  Clinical assessment of the severity of plaque psoriasis
Change in Psoriasis Area and Severity Index from Baseline at 1 Month | After 1 month of treatment.
  Clinical assessment of the severity of plaque psoriasis
Change in Psoriasis Area and Severity Index from Baseline at 2 Months | After 2 months of treatment.
  Clinical assessment of the severity of plaque psoriasis
Change in Psoriasis Area and Severity Index from Baseline at 3 Months | After 3 months of treatment.
  Clinical assessment of the severity of plaque psoriasis

SECONDARY OUTCOMES:
Change in Heart Rate Variability from Baseline at 1 Week | After 1 week of treatment.
  Heart rate variability will be determined from ECG recordings
Change in Heart Rate Variability from Baseline at 1 Month | After 1 month of treatment.
  Heart rate variability will be determined from ECG recordings
Change in Heart Rate Variability from Baseline at 2 Months | After 2 months of treatment.
  Heart rate variability will be determined from ECG recordings
Change in Heart Rate Variability from Baseline at 3 Months | After 3 months of treatment.
  Heart rate variability will be determined from ECG recordings
Change in Plasma Cytokine Levels from Baseline at 1 Week | After 1 week of treatment.
  Plasma concentrations (pg/mL) for 8 different cytokines (GM CSF, IFN-γ, IL-2, IL-4, IL-6, IL-8, IL-10, and TNF-α) will be determined from blood samples.
Change in Plasma Cytokine Levels from Baseline at 1 Month | After 1 month of treatment.
  Plasma concentrations (pg/mL) for 8 different cytokines (GM CSF, IFN-γ, IL-2, IL-4, IL-6, IL-8, IL-10, and TNF-α) will be determined from blood samples.
Change in Plasma Cytokine Levels from Baseline at 2 Months | After 2 months of treatment.
  Plasma concentrations (pg/mL) for 8 different cytokines (GM CSF, IFN-γ, IL-2, IL-4, IL-6, IL-8, IL-10, and TNF-α) will be determined from blood samples.
Change in Plasma Cytokine Levels from Baseline at 3 Months | After 3 months of treatment.
  Plasma concentrations (pg/mL) for 8 different cytokines (GM CSF, IFN-γ, IL-2, IL-4, IL-6, IL-8, IL-10, and TNF-α) will be determined from blood samples.
Change from baseline in cytokine release from cultured leukocytes at 1 week | After 1 week of treatment.
  Cytokine concentrations (pg/mL) for 8 different cytokines (GM CSF, IFN-γ, IL-2, IL-4, IL-6, IL-8, IL-10, and TNF-α) will be measured in supernatant from LPS-stimulated leukocyte cultures.
Change from baseline in cytokine release from cultured leukocytes at 1 month | After 1 month of treatment.
  Cytokine concentrations (pg/mL) for 8 different cytokines (GM CSF, IFN-γ, IL-2, IL-4, IL-6, IL-8, IL-10, and TNF-α) will be measured in supernatant from LPS-stimulated leukocyte cultures.
Change from baseline in cytokine release from cultured leukocytes at 2 months | After 2 months of treatment.
  Cytokine concentrations (pg/mL) for 8 different cytokines (GM CSF, IFN-γ, IL-2, IL-4, IL-6, IL-8, IL-10, and TNF-α) will be measured in supernatant from LPS-stimulated leukocyte cultures.
Change from baseline in cytokine release from cultured leukocytes at 3 months | After 3 months of treatment.
  Cytokine concentrations (pg/mL) for 8 different cytokines (GM CSF, IFN-γ, IL-2, IL-4, IL-6, IL-8, IL-10, and TNF-α) will be measured in supernatant from LPS-stimulated leukocyte cultures.

CONTACTS AND LOCATIONS:
Overall Officials: Harald M Stauss, MD, PhD, Principal Investigator — Burrell College of Osteopathic Medicine
Locations (1):
- Burrell College of Osteopathic Medicine, Las Cruces, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No